CLINICAL TRIAL: NCT05454774
Title: A Clinical Study of AAV Vector Expressing Human Coagulation Factor FVIII Gene Therapy for Hemophilia A
Brief Title: A Study of FVIII Gene Therapy for Hemophilia A
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022019
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; gene therapy; Adeno-Associated Virus
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM 002 (Experimental): 1×10^13 vg/kg, Single-dose treatment.
  Interventions: Genetic: Single dose intravenous injection of BBM 002

INTERVENTIONS:
Genetic: Single dose intravenous injection of BBM 002 — Single dose intravenous infusion of BBM 002, an adeno-associated virus (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor VIII (hFVIII) transgene in liver. The dose of BBM 002 will be 1×10^13 vg/ kg

SUMMARY:
This is a single-arm, open-label, clinical study to evaluate the safety, tolerability of BBM 002 injection in Hemophilia A subjects with residual factor VIII (FVIII) levels ≤2 International unit per deciliter (IU/dl) .

BBM 002 injection is an adeno-associated virus (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor VIII (hFVIII) transgene and raises circulating levels of endogenous FVIII.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully aware of the purpose, nature, methods and possible adverse reactions of the trial and voluntarily sign informed consent.
2. Males ≥ 18 years of age.
3. Have hemophilia A with ≤2 IU/dL (≤2 %) endogenous FVIII activity levels.
4. Have had ≥150 prior exposure days (EDs) to any recombinant and/or plasma-derived FVIII protein products.
5. Have had bleeding events and/or infusions with FVIII protein products (including recombination and plasma source) during the last 12 weeks documented in the subjects' medical records.
6. Have no prior history of hypersensitivity or anaphylaxis associated with any FVIII or IV immunoglobulin administration.
7. Have no FVIII inhibitor. (eg <0.6BU/ml Bethesda Units; or the patient's FVIII inhibitor titer was detected <0.6BU/ml in 2 consecutive times within 1-4 weeks using Bethesda method or Nijmegen method), or no prior medical history of FVIII inhibitor after 150 EDs of FVIII products; no clinical signs or symptoms of decreased response to FVIII products infusion.
8. Agree to use a reliable barrier contraception method from the beginning of signing the informed consent to 52 weeks after BBM002 infusion.
9. Compliance is good, patients and their families have the will of 'gene therapy' clinical trials.

Exclusion Criteria:

1. Being positive for hepatitis B surface antigen (HBsAg) or hepatitis B virus-DNA (HBV-DNA). Being positive for hepatitis C virus antibody (HCV-Ab) or hepatitis C virus RNA (HCV-RNA).
2. Currently on antiviral therapy for hepatitis B or C.
3. Patients with coagulation disorders in addition to hemophilia A.
4. Use of any other systematic immunosuppressant other than glucocorticoids within 30 days prior to enrollment.
5. Patients with vaccination history within 30 days prior to screening.
6. Have potential liver diseases, such as previous diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy or liver fibrosis (fibrosis stage ≥ 3); nodules or cysts were found by B ultrasound, or elevated alpha-fetoprotein was detected by laboratory tests. Subjects who are not eligible for the study if the abnormalities are clinically significant by researchers.
7. Patients with known planned major surgery schedule during the 52-week study period aren't eligible.
8. Have participated in a previous gene therapy research trial before screening, or in a clinical study with an investigational drug within 5 half-life of the investigational product, whichever is longer.
9. Have alcohol or drug dependence, or cannot stop drinking throughout the study. 10.Any concurrent clinically significant major disease or condition that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | 10 weeks
  To access the numbers of DLT events determined by the Safety Data Review Committee (SRC) within 10 weeks after administration
The incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 52weeks
  To assess the safety of BBM 002 Injection by TEAEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Chair — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No